CLINICAL TRIAL: NCT02702947
Title: EFFICACY EVALUATION OF PRUNUS DOMESTICA EXTRACT ON BENIGN PROSTATE HYPERPLASIA (BPH): An Add on Study
Brief Title: Efficacy of Prunus Domestica Extract in BPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chemical Resources (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CR/ BPH /11/13
Record Dates: First submitted 2015-09-29; First posted 2016-03-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-05

CONDITIONS: BPH
Keywords: BPH; Prunus Domestica extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prunus Domestica (Experimental): Prunus domestica extract capsules, 100mg, BD
  Interventions: Dietary Supplement: Prunus domestica extract

INTERVENTIONS:
Dietary Supplement: Prunus domestica extract — Prosman 1 capsule twice a day
  Other Names: Prosman

SUMMARY:
Benign prostatic hyperplasia (BPH) is a nonmalignant enlargement of the prostate Prunus domestica bark contains three groups of active constituents: phytosterols (including beta-sitosterol), pentacyclic triterpenoids (including ursolic and oleaic acids) and ferulic esters of long-chain fatty alcohols (including ferulic esters of docosanol and tetracosanol).

The phytosterols, particularly beta-sitosterol, are found in numerous plants and are anti-inflammatory, inhibiting the synthesis of prostaglandins. Beta-sitosterol has been shown to be useful in cases of BPH by helping to reduce the normally elevated levels of prostaglandins in these patients.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a nonmalignant enlargement of the prostate. Symptoms related to BPH are one of the most common problems in older men. Histological evidence of BPH is found in more than is approximately 10% for men in their 30s, 20% for men in their 40s, reaches 50% to 60% for men in their 60s, and is 80% to 90% for men in their 70s and 80s. The majority of men over the age of 60 are considered to have urinary symptoms attributable to BPH.

The proliferative disorder resulting in BPH affects both the stromal and the epithelial portions of the prostate. The enlarging prostate results in the progressive occlusion of the proximal urethra and can result in both obstructive and irritative urinary tract symptoms.

The preferred medical treatment for many men with symptomatic benign prostatic hyperplasia is either an alpha-adrenergic-receptor antagonist (alpha-blocker), which reduces smooth-muscle tone in the prostate, and bladder neck, or a 5α-reductase inhibitor, which reduces prostate volume by inducing epithelial atrophy. These drugs have side effects including:-dizziness, fatigue, hypotension, headache, insomnia, gynecomastia, and retrograde ejaculation.

The use of plants and herbs for medicinal purposes (phytotherapy) including treatment of BPH symptoms has been growing steadily in most countries. Usage of plant extracts is common in many countries of the world and is increasing in the United States. Phytotherapeutic agents represent nearly half of the medications dispensed for BPH in Italy, compared with 5% for alpha blockers and 5% for 5-alpha reductase inhibitors. In Germany and Austria, phytotherapy is the first-line treatment for mild to moderate urinary obstructive symptoms and represents > 90% of all drugs prescribed for the treatment of BPH. In the United States their use has also markedly increased, they are readily available as nonprescription dietary supplements and are often recommended in "natural health food stores or books" for self treatment of BPH symptoms.

Prunus domestica, or European plum, is a small deciduous tree in the Rosaceae (rose) family that is an ancient domesticated species, known only in cultivation. It is now cultivated in temperate areas worldwide for its fruit.

Mechanism of action The bark contains three groups of active constituents: phytosterols (including beta-sitosterol), pentacyclic triterpenoids (including ursolic and oleaic acids) and ferulic esters of long-chain fatty alcohols (including ferulic esters of docosanol and tetracosanol).

The phytosterols, particularly beta-sitosterol, are found in numerous plants and are anti-inflammatory, inhibiting the synthesis of prostaglandins. Beta-sitosterol has been shown to be useful in cases of BPH by helping to reduce the normally elevated levels of prostaglandins in these patients. The elimination of the excess blood and vasal congestion helps reduce the size of prostate adenomas. The pentacyclic triterpenoids also help inhibit inflammation by blocking enzymatic activity. They are effective anti-edema agents and also help increase the integrity of small veins and capillaries. The third active group, the ferulic esters of long-chain fatty acids, act by inhibiting the absorption and metabolism of cholesterol. BPH and other cases of enlarged prostates are characterized by containing abnormally high levels of cholesterol. Plant efficacy was determined by measuring the effects of the herb on numerous parameters, including dysuria, nycturia, frequent urination, abdominal heaviness, residual urine, voiding volume, prostate volume, and peak flow. Consumption of P.Domestica resulted in significant amelioration of symptoms, reduction in prostate size, and clearance of bladder neck urethral obstruction.

Different studies suggest that these phytochemicals appear to work synergistically to improve the symptoms of BPH. However, the most bioactive phytochemicals in pygeum are the phytosterols. Therefore, these components of pygeum extract are believed to exert the most important therapeutic effect in the treatment of BPH.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years
* Only Male included
* Has suffered from symptoms of BPH for at least the 6 months before Screening.
* Has a prostate volume ≥ 20 mL and ≤ 70 mL as assessed by ultrasound
* Has an IPSS ≥ 8 at Screening and Baseline
* Patients willing to give informed consent in writing

Exclusion Criteria:

* Neurogenic bladder dysfunction
* Has bladder neck contracture or urethral stricture
* Has acute or chronic prostatitis or urinary tract infection
* Has a history of, prostate cancer or carcinoma of the prostate suspected on digital rectal exam.
* Participation in any other clinical trial with in the last 30 days
* Has resting systolic blood pressure (BP) > 160 mmHg or < 90 mmHg, or diastolic BP > 90 mmHg or < 60 mmHg at Screening.
* Urine flow< 5mls/sec.
* Use of any other herbal medications for treatment of BPH, associated symptoms and Erectile Dysfunction in past 1 month.
* Has hematuria of unknown etiology.
* Previous radiotherapy

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Reduction in prostate volume | 12 weeks

SECONDARY OUTCOMES:
Improvement in urinary flow parameters | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Satyanarayan sankhwar, M.S., M.Ch., Principal Investigator — King George's Medical University, Lucknow, UP, India; Dr. Narsingh Verma, M.D., Principal Investigator — King George's Medical University, Lucknow, UP, India
Locations (1):
- Department of Urology, King George's Medical University, Lucknow, UP, India, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roehrborn CG. Benign prostatic hyperplasia: an overview. Rev Urol. 2005;7 Suppl 9(Suppl 9):S3-S14. PMID 16985902
- See also: Phytotherapeutic agents in the treatment of benign prostatic hyperplasia — http://link.springer.com/article/10.1007%2Fs11934-000-0044-y#page-1